CLINICAL TRIAL: NCT04575818
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of GLPG4059 in Adult, Healthy, Male Subjects
Brief Title: A Study in Healthy Male Volunteers Investigating the Safety, Absorption and Elimination of Single Doses of GLPG4059
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development of compound has been stopped
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG4059-CL-101; 2020-000036-22 (EudraCT Number)
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part 1 (SAD) is randomized, double-blind, placebo-controlled; Part 2 (FE and rBA) is randomized, open-label.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- GLPG4059 SAD (Experimental): Single doses of GLPG4059 at up to 6 dose levels in ascending order
  Interventions: Drug: GLPG4059 oral suspension
- Placebo SAD (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo
- GLPG4059 rBA/FE oral suspension fasted (Experimental): Single dose of GLPG4059 in fasted state
  Interventions: Drug: GLPG4059 oral suspension
- GLPG4059 rBA/FE tablet fed (Experimental): Single dose of GLPG4059 in fed state
  Interventions: Drug: GLPG4059 tablet
- GLPG4059 rBA/FE tablet fasted (Experimental): Single dose of GLPG4059 in fasted state
  Interventions: Drug: GLPG4059 tablet

INTERVENTIONS:
Drug: GLPG4059 oral suspension — GLPG4059 for oral administration
  Arms: GLPG4059 SAD; GLPG4059 rBA/FE oral suspension fasted
Drug: Placebo — Placebo oral suspension
  Arms: Placebo SAD
Drug: GLPG4059 tablet — GLPG4059 for oral administration
  Arms: GLPG4059 rBA/FE tablet fasted; GLPG4059 rBA/FE tablet fed

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of GLPG4059 in healthy volunteers after single oral administrations of GLPG4059 (SAD), compared to placebo (part 1). The effect of food (FE) (high-fat, high calorie) on the pharmacokinetics and relative bioavailability (rBA) of GLPG4059 will be assessed (part 2).

ELIGIBILITY:
Inclusion Criteria:

* Male between 18-54 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18-30 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and fasting clinical laboratory safety tests, available at screening and prior to randomization. ECG and vital signs parameters must be within the normal ranges. Bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be no greater than 1.5x upper limit of normal (ULN). Fasting plasma glucose must be <6.99 mmol/L, fasting defined as no caloric intake for at least 8 hours and hemoglobin A1c (HbA1c) <6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is national glycohemoglobin standardization program (NGSP) certified and standardized to the diabetes control and complications trial (DCCT) assay. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to Investigational Medicinal Product (IMP) ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the IMP.

This list only contains the key exclusion criteria.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations | From screening through study completion, an average of 7 months
  To evaluate the safety and tolerability of single ascending oral doses of GLPG4059, in adult, healthy, male subjects compared with placebo.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG4059 | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of single ascending oral doses of GLPG4059, in adult, healthy, male subjects.
Area under curve (AUC) of GLPG4059 | Between Day 1 pre-dose and Day 4
  To evaluate the PK of single ascending oral doses of GLPG4059, in adult, healthy, male subjects
Terminal elimination half-life (t1/2) of GLPG4059 | Between Day 1 pre-dose and Day 4
  To evaluate the PK of single ascending oral doses of GLPG4059, in adult, healthy, male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No